CLINICAL TRIAL: NCT05606159
Title: A Randomized, Double-blind, Placebo-controlled Clinical Trial to Evaluate the Tolerability and Effect of Bacillus Velezensis DSM 33864 on the Reduction of Risk of Recurrent Clostridioides Difficile Infection (rCDI) in Adults With a History of rCDI
Brief Title: Bacillus Velezensis DSM 33864 for Reduction of the Risk of Recurrent Clostridioides Difficile Infections
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Research Project closed
Sponsor: Novozymes A/S (Industry)
Collaborators: Estimates OY (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: NZ-GHCD-2021-06
Record Dates: First submitted 2022-08-09; First posted 2022-11-04 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Clostridium Difficile Infection Recurrence
Keywords: Probiotic; Gastrointestinal Microbiota; C. difficile; Dietary supplement
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled multicenter clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bacillus velezensis DSM 33864 (Experimental): This arm will receive a single strain probiotic capsule containing Bacillus velezensis DSM 33864.
  The probiotic will be taken orally, once a day, for 8 weeks.
  Interventions: Dietary Supplement: Bacillus velezensis DSM 33864
- Placebo control group (Placebo Comparator): A placebo capsule containing microcrystalline cellulose will be taken orally, once a day, for 8 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Bacillus velezensis DSM 33864 — 1 probiotic capsule to be taken orally once a day, with breakfast, once a day for 8 weeks.
  Other Names: Probiotic
  Arms: Bacillus velezensis DSM 33864
Dietary Supplement: Placebo — 1 microcrystalline cellulose-containing placebo capsule to be taken orally once a day with breakfast, for 8 weeks.
  Arms: Placebo control group

SUMMARY:
The purpose of this study is to determine whether a single strain capsulated probiotic, when used after standard C. difficile antibiotic therapy, is effective in reducing the risk of infection recurrence mediated by a decrease in colonization by toxigenic C. difficile. This study will include adults with a history of two episodes of C. difficile infection (CDI).

DETAILED DESCRIPTION:
The goal of this multi-center randomized double-blinded placebo-controlled trial is to evaluate the tolerability and effect of a probiotic dietary supplement on the reduction of the risk of recurrent C. difficile infection in adults who have experienced two previous C. difficile infection episodes.

The main aim of this study is to assess the effect of a probiotic dietary supplement on the colonization (cell counts) of C. difficile over time and also to assess the correlation between level of C. difficile colonization and recurrence of CDI.

Approximately, 104 research subjects will be randomized into two arms and will use either one capsule daily of the probiotic supplement or placebo once daily with breakfast, for 8 weeks. All outcomes will be compared across the supplementation and placebo arm.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ≥ 18 years old
2. Medical record documentation of second or subsequent recurrent CDI episode, and received standard-of-care oral antibiotic therapy completed no more than 5 days prior date of enrollment.
3. Able to provide signed and dated informed consent or assent
4. Able to provide blood and fecal specimens

Exclusion Criteria:

1. Current episode of CDI or delayed symptom resolution from previous reoccurrence (second episode), according to the physical exam and investigator assessment
2. Pregnancy or breastfeeding
3. Subjects presenting with active diarrhea (3 or more stools per 24-hour period) and within Bristol stool scale range of 5-7
4. Taking dietary supplement or therapeutic intervention which could significantly affect parameter(s) followed during the study (fibers, probiotics, prebiotics, symbiotic) according to the investigator or stopped in a too short period before the V1 visit (< 4 weeks)
5. Previous reaction, including anaphylaxis, to any substance in composition of the study product
6. Active, non-controlled intestinal disease such as Crohn's Disease, ulcerative colitis; celiac disease, or other chronic diarrheal illness
7. Patients with active Pancreatitis
8. Ostomized subjects, parenteral nutrition users
9. Under immunosuppressive therapy or any health condition causing immunosuppression (including active hematological malignancies, acquired immune deficiency syndrome (AIDS), recent solid organ transplant (within 90 days),under treatment for rejection
10. For women: Non menopausal with the same reliable contraception since at least 3 cycles before the beginning of the study and agreeing to keep it during the entire duration of the study or menopausal without or with hormone replacement therapy (estrogenic replacement therapy begun from less than 3 months excluded);
11. Pregnant or lactating women or intending to become pregnant within 3 months ahead

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-11 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
C. difficile colonization | 8 weeks
  Change in colonization (counts) of toxigenic C. difficile from baseline to 8 weeks determined by quantitative PCR

SECONDARY OUTCOMES:
C. difficile colonization | 4 weeks
  Change in colonization (counts) of toxigenic C. difficile determined by quantitative PCR
C.difficile colonization | 12 weeks
  Change in colonization (counts) of toxigenic C.difficile determined by quantitative PCR
Presence and levels of C. difficile toxin in fecal samples | 12 weeks
  Change in concentration of C. difficile Toxin A or B levels in fecal samples from baseline to week 4, week 8 and week 12 determined by enzyme immune assay method (EIA)
Quality of life assessment | 12 weeks
  Change in average health-related quality of life scores at baseline, week 8 and 12, determined by EQ-5D-5L questionnaire
Reduction of the risk of rCDI | 8 weeks
  Incidence of rCDI defined as an episode of diarrhea onset described by three or more unformed stools per 24 h as measured by the Bristol stool chart (types 5 to 7), and positive toxin assay result for C. difficile.
Reduction of the risk of rCDI | 4 weeks
  Incidence of rCDI defined as an episode of diarrhea onset described by three or more unformed stools per 24 h as measured by the Bristol stool chart (types 5 to 7), and positive toxin assay result for C. difficile.

OTHER OUTCOMES:
Incidence of adverse events | 12 weeks
  Incidence of adverse events from baseline to 12 weeks
Changes in hemoglobin concentration | 12 weeks
  Changes in hemoglobin concentration from baseline to 12 weeks determined by standard Full Blood Count (FBC) test
Changes in blood platelet levels | 12 weeks
  Changes in blood platelet levels from baseline to 12 weeks determined by standard Full Blood Count (FBC) test
Changes in blood C-reactive protein (CRP) levels | 12 weeks
  Changes in C-reactive levels from baseline to 12 weeks determined by standard blood CRP test
Changes in blood glucose levels | 12 weeks
  Changes in blood glucose from baseline to 12 weeks determined by standard blood chemistry panel test
Changes in blood urea nitrogen (BUN) levels | 12 weeks
  Changes in blood urea nitrogen levels from baseline to 12 weeks determined by standard blood chemistry panel test
Changes in blood creatinine levels | 12 weeks
  Changes in blood creatinine levels from baseline to 12 weeks determined by standard blood chemistry panel test
Changes in blood calcium levels | 12 weeks
  Changes in blood calcium levels from baseline to 12 weeks determined by standard blood chemistry panel test
Incidence of any diarrhea determined by the Bristol Stool Scale (score range 5-7) | 12 weeks
  Incidence of any diarrhea determined by the Bristol Stool Scale (score range 5-7)
Incidence of gastrointestinal pain or discomfort determined by GSRS questionnaire | 12 weeks
  Incidence of gastrointestinal pain or discomfort determined by GSRS questionnaire
Intestinal microbiome diversity including functional and resistome genes | 8 weeks
  Change in intestinal microbiome composition assessed from fecal samples using Deep Shotgun sequencing method
Change in intestinal bile acid levels | 12 weeks
  Change in bile acids assessed from fecal samples by UPLC-MS
Change in intestinal short-chain fatty-acid levels | 12 weeks
  Change in short chain fatty acids assessed from fecal samples by GC-MS
Recovery rate of Bacillus velezensis assessed from fecal samples | 12 weeks
  Recovery rate of probiotic Bacillus velezensis DSM33864 in fecal samples, determined by qPCR method

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Sims, PhD, Principal Investigator — Beaumont Hospital, Royal Oak. Michigan
Locations (1):
- Beaumont Hospital, Royal Oak, Michigan, United States

IPD SHARING:
Plan to Share IPD: No